CLINICAL TRIAL: NCT07198503
Title: Study on Carotenoid-Based Instrumental Index
Status: Recruiting | Type: Observational
Sponsor: ChinaNorm (Industry)
Collaborators: Nu Skin Enterprises (Industry)
Responsible Party: Sponsor
Other Study IDs: W25002001
Record Dates: First submitted 2025-09-12; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Skin Carotenoid Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chinese citizens aged 18-50: The study sample was selected to be as evenly distributed as possible in terms of age and gender.
- Chinese citizens aged ≥50: The study sample was selected to be as evenly distributed as possible in terms of age and gender.

SUMMARY:
Nu Skin (China) Daily-Use&Health Products Co.,Ltd. has developed biophotonic scanners based on Raman spectroscopy, which measures skin carotenoid levels through hand skin scanning. In this study, the new Prysm device, which adopts new technology in a lower cost and more portable form, was used to measure skin carotenoid levels in a population, and the relationships between these levels and dietary habits and lifestyle factors were analyzed. The collected data included basic demographic information such as age, gender, smoking status, use of health products or nutritional supplements, and exercise habits, as well as physiological indicators such as BMI and body fat percentage. Subjective assessments were also obtained, including questionnaires on diet, skin condition, physical health, lifestyle, psychological status, and memory performance, alongside skin image analyses capturing parameters such as ITA°, L*, a*, b*, glossiness, erythema, and pigmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese individuals of Asian ethnicity aged 18 years or older.
2. Basic proficiency in reading and writing Chinese, sufficient to independently complete questionnaires.
3. Voluntary participation with signed informed consent.
4. Willingness to comply with all assessment requirements.

Exclusion Criteria:

1. Presence of open facial lesions, prominent scars, or visible acne marks.
2. Currently planning pregnancy, pregnant, or breastfeeding.
3. Ongoing treatment for acute or severe medical conditions.
4. Significant impairments affecting cognitive or behavioral abilities.
5. Other medical reasons identified by experts or professionals that may interfere with the assessment results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese individuals of Asian ethnicity aged 18 years or above.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-06 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Skin Carotenoid Index | At a single Day 1 visit after enrollment
  The Prysm device utilizing hyperspectral absorption technology and the S3 device utilizing Raman spectroscopy technology, was used to measure the skin carotenoid index on subjects' fingers.
Body Mass Index (BMI) | At a single Day 1 visit after enrollment
  BMI is derived from the subjects' measured height and weight.
Body Fat Percentage (BF%) | At a single Day 1 visit after enrollment
Demographic Information | At a single Day 1 visit after enrollment
  Including basic information such as gender, age, smoking status, use of health products or nutritional supplements, exercise habits.
Dietary Intake | At a single Day 1 visit after enrollment
  Subjects' dietary intake during the previous month was evaluated using Food Frequency Questionnaire - 25 (FFQ-25).
Fitzpatrick Skin Type | At a single Day 1 visit after enrollment
Skin Condition Self-Assessment | At a single Day 1 visit after enrollment
  Subjects evaluated their skin condition during the previous month using a self-assessment questionnaire, covering dimensions such as photodamage, skin brightness, skin radiance, etc. Each dimension is scored from 0 to 9, with higher scores indicating better skin condition.
The score of 36-Item Short Form Survey (SF-36) | At a single Day 1 visit after enrollment
  It consists of 9 different dimensions: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), Mental Health (MH), Reported Health Transition (HT). Each dimension is scored from 0 to 100, higher scores reflect better health, functionality, and quality of life.
Frequency of Physical Illness Symptoms | At a single Day 1 visit after enrollment
  Subjects' immune function over the past year was evaluated using a questionnaire that collected the frequency of symptoms, including colds, influenza, allergies, etc. The total score ranges from 0 to 28, higher scores are associated with poorer immune function.
Gastrointestinal Discomfort Symptoms | At a single Day 1 visit after enrollment
  Subjects' gastrointestinal discomfort over the past month, including symptoms such as abdominal pain and bloating, was assessed using a questionnaire. The total score ranges from 20 to 100, and higher scores reflect more severe symptoms of gastrointestinal discomfort.
Population-Based Visual Fatigue Scale Score | At a single Day 1 visit after enrollment
  The questionnaire comprises 5 ocular symptoms (such as 'discomfort around the eyes', 'dryness of the eyes', etc.) and 6 visual and systemic symptoms (such as 'eye discomfort caused by screen brightness', 'anxiety associated with eye discomfort', etc.). The total score ranges from 0 to 44, higher scores reflect greater symptom severity.
Traditional Chinese Medicine (TCM) Constitution Classification | At a single Day 1 visit after enrollment
  Subjects' body constitution was evaluated and categorized based on the Traditional Chinese Medicine Constitution Classification and Determination Self-Assessment Form, following the standards of the China Association of Chinese Medicine. For each constitution classification, scores range from 0 to 100, and higher scores indicate greater alignment with specific body constitution.
Brief Resilience Scale (BRS) Score | At a single Day 1 visit after enrollment
  The BRS score is calculated by summing averaging the scores of all the six items, which ranges from 1 to 5. A higher average indicates greater psychological resilience, while a lower average indicates lower psychological resilience.
Multifactorial Memory Questionnaire (MMQ) Score | At a single Day 1 visit after enrollment
  It consists of three subscales: How I Feel About My Memory (scores range from 0 to 72), Memory Mistakes (scores range from 0 to 80) and Use of Memory Strategies (scores range from 0 to 68). A higher score indicates better memory.
Facial image analysis | At a single Day 1 visit after enrollment
  Including red area ratio, number and area ratio of color spots, L, a, b, and ITA °.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided